CLINICAL TRIAL: NCT03814525
Title: Evaluation of Photobiomodulation Effects on Pain, Edema, Paresthesia and Bone Regeneration After Maxillar Surgical Disjunction: Double Blind, Randomized and Controlled Clinical Trial
Brief Title: Photobiomodulation Effects on Pain, Edema, Paresthesia and Bone Regeneration After Maxillar Surgical Disjunction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Eduardo
Record Dates: First submitted 2019-01-18; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Maxillary Diseases
MeSH Terms: conditions — Maxillary Diseases | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The pre and postoperative evaluations will be done by two examiners who will not be aware of the group in which each patient is allocated. The information that will be obtained in the evaluations will be noted in the clinical evaluation card. Participants will not be aware of whether or not they have received the FBM, since the person responsible for the application will position the equipment in the irradiation locations in all participants and will only trigger the light when and where predicted in the specific experimental group. The characteristic sound of the device will be triggered by recording in the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (Active Comparator): PBM will be applied after the surgeries with extra and intraoral LED devices. The LED plates speed up the treatment as they deliver all the energy at once, having the advantage of radiating several points at the same time. The applications of both will occur in the following experimental periods after the end of the surgeries: immediate postoperative, 1, 2, 7, 14, 30, 60 and 90 days.
  Interventions: Radiation: Photobiomodulation
- Control group (Placebo Comparator): Participants will be attended in the same way as the PBM group. The person who is responsible for the application of the PMB will simulate the irradiations by positioning the devices in the same locations described for the PBM group, but the equipment will be kept off.
  Interventions: Radiation: Placebo Photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation — PBM will be applied with extra and intraoral LED devices. The LED plates speed up the treatment as they deliver all the energy at once, having the advantage of radiating several points at the same time. The applications of both will occur in the following experimental periods after the end of the surgeries: immediate postoperative, 1, 2, 7, 14, 30, 60 and 90 days.
  Arms: Photobiomodulation group
Radiation: Placebo Photobiomodulation — The person responsible for applying the PBM will simulate the irradiation by positioning the devices in the same locations described for the PBM group, but the equipment will be kept off
  Arms: Control group

SUMMARY:
The objective of the present study will be to evaluate the efficacy of photobiomodulation (PBM) with LED in pain control, facial edema, paresthesia, bone repair and quality of life arising after maxillar surgical disjunction (MSD). A randomized, double-blind, placebo-controlled clinical trial involving 72 participants aged 18 to 45 years, who search the Service of Oral Maxillofacial Surgery and Traumatology of the Mandaqui Hospital Complex to undergo MSD, attend to the eligibility criteria and agree to participate. Surgeries will be conducted by three oral maxillofacial surgeons who will perform all surgical procedures, two examiners (who will perform pre and post-surgical evaluations, blinded to the experimental group) and another researcher who will perform the LED application. Before the surgeries, facial measures, radiographic examinations, tests of facial and oral sensitivity and the evaluation of the level of anxiety of all the participants will be carried out. Immediately after the surgeries, the participant will be inserted into the placebo group or the LED group, according to block randomization defined previously. In the LED group, the participants will receive PBM with an extraoral device (660 and 850 nm with 6J per point) and an intraoral one (660 nm with 2J per point) and in the control group the participants will be attended in the same way, but with the LED devices kept off. The applications will be in the immediate postoperative period, 1, 2, 7, 14, 30, 60, 90 and 120 days after the end of the surgeries, when the evaluations will also be performed. Facial measurements, extra and intraoral sensitivity, pain and bone repair will be evaluated. Secondarily, the data regarding the occurrence of headache; otalgia; nausea; bruise; nasolacrimation; epistaxis; dysphagia; systemic and superficial temperature in the operated region; use of analgesics and anti-inflammatories; anxiety and impact of oral health on the participants' quality of life will be computed.

ELIGIBILITY:
Inclusion Criteria:

* Transverse maxillary deficiency ˃ of 5 mm with bilateral posterior crossbite and indication for surgical maxillary disjunction.
* Agree to participate in the study after reading and signing the Term of Consent for Participation in Clinical Research.

Exclusion Criteria:

* Transverse maxilla deficiency, with unilateral posterior crossbite.
* Local or systemic alterations that contraindicate surgical intervention or hinder the postoperative period.
* Smokers.
* Display photo sensitivity history.
* Possess systemic diseases, chronic pain or neurological and psychiatric disorders.
* Have been using anti-inflammatories, analgesics or bisphosphonates in the past 15 days.
* Pregnant.
* Breastfeeding.
* Participants who present any type of complication during surgery (hemorrhage, operative difficulty), as these cases will not be in the expected pattern for these surgeries. These data will not be part of the statistical analysis but will be described and discussed, as well as possible adverse effects.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | After 1, 2, 7 and 14 days of surgeries.
  A Visual Analog Scale (VAS) will be printed on the patient evaluation form and the subjects will be instructed by the evaluator to mark a point in the line of 10 cm, indicating the intensity of their pain after 1,2, 7 and 14 days of the surgeries. For the NRS-101 scale, the evaluators will ask patients to assign a number between 0 (no pain) and 100 (worst possible pain) that best represents the pain they are currently experiencing after 1, 2, 7 and 14 days of surgeries.
Change in Edema | After 1, 2, 7 and 14 days of surgeries.
  Using a flexible plastic millimeter tape (0.5mm precision), five facial measurements will be taken corresponding to the distances between the points listed below as described by Ristow et al. (2013).
  Line A - posterior tragus point to the most lateral point of the labial commissure Line B - tragus posterior point to pogonium Line C - posterior tragus point to the lateral corner of the eye Line D - lateral corner of eye to lowest point of jaw angle Line E - lower point of the angle of the mandible (gonio) to the middle of the nasal bone
Change in intra and extraoral sensitivity | After 7, 30, 60, 90 and 120 days of surgeries.
  The evaluation of extra and intraoral sensitivity will be performed in 6 regions: below the lower eyelid, cheek, nose wing, upper lip, oral buccal mucosa and oral palatal mucosa on both sides. The tests will be performed sequentially, with a 2 to 3 minute interval between each. The participant will receive instructions on the tests that will be initially performed on the back of his hand so he can become familiar.
Change in postoperative bone repair | After 30, 60, 90 and 120 days of surgeries.
  The optical density (OD) of the alveolar bone in the anterior region of the palatine suture, in each experimental period, will be calculated and compared with that obtained in the preoperative radiographic examination.

SECONDARY OUTCOMES:
Change in temperature | After 1, 2, 7 and 14 days of surgeries.
  The temperature will be measured locally (on both sides) and systemically. Local measurements will be measured using an infrared digital thermometer in the right and left cheek region and anterior nasal spine. The systemic temperature will be measured in the frontal region of the patient in the median position 3 cm above the glabella.
Presence of headache | After 1, 2, 7 and 14 days of surgeries.
  Patients will answer yes or not, to indicate whether they had headaches in the examined periods.
Presence of bruises | After 1, 2, 7 and 14 days of surgeries.
  The presence of hematoma/ecchymosis will be evaluated by measuring the largest diameter of the colorimetric changes on the right and left side. The measure will be performed by the examiners who will classify the occurrence of this result into four categories: 1) none; 2) larger diameter smaller than 4 cm; 3) larger diameter between 4 and 10 cm, and 4) larger diameter greater than 10 cm.
Presence of otalgia | After 1, 2, 7 and 14 days of surgeries.
  Patients will answer yes or not, to indicate whether they had otalgia in the examined periods.
Presence of nausea | After 1, 2, 7 and 14 days of surgeries.
  Patients will answer yes or not, to indicate whether they had nausea in the examined periods.
Presence of nasolacrimation | After 1, 2, 7 and 14 days of surgeries.
  Patients will answer yes or not, to indicate whether they had nasolacrimation in the examined periods.
Presence of nose bleeding | After 1, 2, 7 and 14 days of surgeries.
  Patients will answer yes or not, to indicate whether they had nose bleeding in the examined periods.
Presence of dysphagia | After 7 and 30 days of surgeries.
  The evaluation of dysphagia will be performed after 7 and 30 days by questioning and classification on a numerical scale in which:
  (0) total absence of dysphagia;
  1. dysphagia to solid foods
  2. dysphagia to any liquid or solid food
Postoperative quality of life | After 7 and 30 days of surgeries.
  Patients will answer yes or no to the following questions:
  1. Are you maintaining your social activities normally?
  2. Are you working / studying normally?
  3. Are you maintaining your normal diet?
  4. Do you have difficulty swallowing because of the surgery?
  5. Do you have difficulty in tasting food?
  6. Can you chew on the sides?
  7. Do you have trouble sleeping because of the surgery?
  8. Did you have trouble speaking because of the surgery?
  9. Has your appearance changed because of the surgery?
  10. Do you feel sick from the surgery?

CONTACTS AND LOCATIONS:
Locations (1):
- Conjunto Hospitalar do Mandaqui, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] da Fonseca EV, Bussadori SK, da Silva Martinho LFC, de Sousa Melo MC, de Andrade FL, Goncalves MLL, Mesquita-Ferrari RA, Horliana ACRT, Fernandes KPS. Evaluation of photobiomodulation effects on pain, edema, paresthesia, and bone regeneration after surgically assisted rapid maxillary expansion: Study protocol for a randomized, controlled, and double blind clinical trial. Medicine (Baltimore). 2019 Nov;98(48):e17756. doi: 10.1097/MD.0000000000017756. PMID 31770194